CLINICAL TRIAL: NCT02812030
Title: Aflibercept for Retinopathy in the Real World (ARRoW) Study: Evaluation of Anti-VEGF Treatment for Diabetic Macular Oedema
Brief Title: Aflibercept for Retinopathy in the Real World
Acronym: ARRoW
Status: Withdrawn | Type: Observational
Why Stopped: Superceded by a larger trial by the pharmaceutical company
Sponsor: Timothy Jones (Other)
Collaborators: University Hospitals Bristol and Weston NHS Foundation Trust (Other); Gloucestershire Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor-Investigator, Timothy Jones, Senior Research Associate, University of Bristol
Organization: University of Bristol (Other)
Other Study IDs: P201
Record Dates: First submitted 2016-06-22; First posted 2016-06-23 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Diabetic Retinopathy
Keywords: Observational Study; aflibercept; Diabetic Retinopathy; Visual Acuity
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- aflibercept in real world: Patients receiving aflibercept for diabetic macular oedema at Bristol Eye Hospital or Gloucestershire Hospitals NHS Foundation Trust
  Interventions: Other: National Eye Institute Visual Functioning Questionnaire

INTERVENTIONS:
Other: National Eye Institute Visual Functioning Questionnaire — Routine treatment plus visual functioning questionnaires
  Other Names: NEIVFQ-25

SUMMARY:
Diabetic retinopathy remains the leading cause of blindness in patients of working age in the Western World, and there is a global epidemic of diabetes. The recommended treatment for diabetic retinopathy involves injection of anti-vascular endothelial growth factor (anti-VEGF) into the eye. Based on two recent clinical trials taking place in the United States, Europe, Japan, and Australia, NICE issued guidance in July 2015 recommending that aflibercept (a particular type of anti-VEGF treatment) should be available on the NHS for patients in whom the central retina of the eye is at least 400 micrometres thick before treatment.

Real-world data can differ significantly from clinical trial data, and it is therefore very important to evaluate the impact of aflibercept in a real world setting, particularly with respect to systemic control, as patients with poor systemic control were excluded from the clinical trials. This study aims to demonstrate the efficacy of aflibercept in a real-world setting, and how this compares to the clinical trial setting.

DETAILED DESCRIPTION:
Participants will receive treatment as usual for diabetic macular oedema at Bristol Eye Hospital (University Hospitals Bristol NHS Foundation Trust) and Gloucestershire Hospitals NHS Foundation Trust. This entails injection of aflibercept into the eye, initially with four monthly doses, then as required with regular monthly assessments. Additionally, patients will be invited to complete standardised visual functioning questionnaires at baseline and roughly 6 and 12 months. Patients will be followed up for one year for this study, but treatment will continue as necessary beyond the end of the study.

The primary outcome of Best-Corrected Visual Acuity (BCVA) will be assessed at one year and compared to the treatment arm of two recent phase 3 RCTs (VISTA and VIVID). Additional secondary outcomes of retinal thickness, visual functioning, and adverse events will also be collected.

Real world data will be collected from Bristol Eye Hospital and Gloucestershire Hospitals NHS Foundation Trust. Bristol Eye Hospital, as part of the RENOIR HIT, has set up a hub and spoke outreach model to treat patients with diabetic macular oedema, and this service has been running since September 2013. Treatment is performed at one of three outreach sites: South Bristol Community hospital, St Georges medical practice in Worle, and a mobile macular unit currently based at Cribbs Causeway. There are about three to five new patients per month commencing treatment with aflibercept in the Bristol area. In Gloucestershire, treatments are performed at Cheltenham General Hospital, and Gloucester Royal Hospital; we expect an additional two to three new patients per month from these sites.

All patients attending for routine treatment will be invited to take part in the study. In order to detect a clinically significant difference of 5 letters using the Early Treatment of Diabetic Retinopathy Study (ETDRS) protocol, between the real world and the clinical trials, sample size calculations suggest we will need at least 30 new patients to compare to the treatment arm of the clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18+ years
* Eligible for NHS treatment under the auspices of Bristol Eye Hospital (3 outreach locations) or Gloucestershire NHS Foundation trust.
* Diagnosis of centre-involving diabetic macular oedema
* Receiving a first ever treatment of aflibercept in a new eye

Exclusion Criteria:

* Any previous anti-vascular endothelial growth factor (anti-VEGF) treatment in the study eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults receiving their first ever treatment with aflibercept for diabetic macular oedema
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Change in Best-Corrected Visual Acuity (BCVA) | Baseline - 12 months
  Best-corrected visual acuity using a standardised measure involving number of Early Treatment Diabetic Retinopathy Study (ETDRS) letters.

SECONDARY OUTCOMES:
Change in central retinal thickness | Baseline - 12 months
  Central retinal thickness measured using optical coherence tomography
Ocular adverse events | 12 months
  Eye-related adverse events (e.g., endophthalmitis, uveitis, increased intraocular pressure)
Non-ocular adverse events | 12 months
  Non-eye-related adverse events (e.g., death, stroke, TIA)

CONTACTS AND LOCATIONS:
Overall Officials: Clare Bailey, MA, BM, BCh(Oxon), MRCP, Principal Investigator — University Hospitals Bristol and Weston NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Diabetic Retinopathy Clinical Research Network; Wells JA, Glassman AR, Ayala AR, Jampol LM, Aiello LP, Antoszyk AN, Arnold-Bush B, Baker CW, Bressler NM, Browning DJ, Elman MJ, Ferris FL, Friedman SM, Melia M, Pieramici DJ, Sun JK, Beck RW. Aflibercept, bevacizumab, or ranibizumab for diabetic macular edema. N Engl J Med. 2015 Mar 26;372(13):1193-203. doi: 10.1056/NEJMoa1414264. Epub 2015 Feb 18. PMID 25692915
- [Background] Do DV, Nguyen QD, Boyer D, Schmidt-Erfurth U, Brown DM, Vitti R, Berliner AJ, Gao B, Zeitz O, Ruckert R, Schmelter T, Sandbrink R, Heier JS; da Vinci Study Group. One-year outcomes of the da Vinci Study of VEGF Trap-Eye in eyes with diabetic macular edema. Ophthalmology. 2012 Aug;119(8):1658-65. doi: 10.1016/j.ophtha.2012.02.010. Epub 2012 Apr 24. PMID 22537617
- [Background] Korobelnik JF, Do DV, Schmidt-Erfurth U, Boyer DS, Holz FG, Heier JS, Midena E, Kaiser PK, Terasaki H, Marcus DM, Nguyen QD, Jaffe GJ, Slakter JS, Simader C, Soo Y, Schmelter T, Yancopoulos GD, Stahl N, Vitti R, Berliner AJ, Zeitz O, Metzig C, Brown DM. Intravitreal aflibercept for diabetic macular edema. Ophthalmology. 2014 Nov;121(11):2247-54. doi: 10.1016/j.ophtha.2014.05.006. Epub 2014 Jul 8. PMID 25012934